CLINICAL TRIAL: NCT07318662
Title: Efficacy and Safety of HMAs Combined With Venetoclax Versus HMAs Alone in Newly Diagnosed Patients With Intermediate-/High-Risk MDS and CMML : A Retro-prospective, Multicenter Observational Cohort Study
Brief Title: Efficacy and Safety of HMAs Combined With Venetoclax Versus HMAs Alone in ND Int-and H-risk MDS or CMML
Status: Active, not recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Du Xin, professor of medical science, Guangdong Provincial People's Hospital
Other Study IDs: GDPH-2024-MDS-1.2
Record Dates: First submitted 2025-11-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: MDS; CMML
Keywords: MDS; CMML; Venetoclax; Hypomethylating agents
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Venetoclax+HMAs: treatment group, the intervention is the use of Venetoclax(400mg，QD, 1-14d)
  Interventions: Drug: Venetoclax
- Standard treatment(HMAs): The control group，Azacitidine（75mg/m2 ，QD, sc，d1-d7）or Decitabine（15mg/m2, q8h-q12h, d1-d3 or 20mg/m2,qd, d1-d5)

INTERVENTIONS:
Drug: Venetoclax — Previous phase Ib studies have fully demonstrated that venetoclax combined with HMAs is well tolerated in patients with MDS or CMML. Patients treated with VEN/AZA had a higher chance of SCT after remission and a higher survival benefit
  Groups: Venetoclax+HMAs

SUMMARY:
The aim of this study is to observe and analyze the clinical efficacy of Venetoclax+HMAs regimen in the treatment of newly diagnosed higher-risk MDS and CMML cases, and to compare the efficacy of venetoclax +HMAs regimen with that of HMAS regimen alone, in order to provide a normative scheme and basis for clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. MDS or CMML diagnosed by the 2016 or 222 WHO criteria, with a sustained survival of at least 12 weeks;
3. received more than two cycles of Venetoclax plus HMAs or HMAs alone without prior disease specific or allogeneic hematopoietic stem cell therapy (before initiating Venetoclax or HMAs, Medications such as hydroxyurea were allowed to reduce the white-cell count to 1.0×109 per liter or less.) ;
4. bone marrow blast cell count (BM blast > 5%) or IPSS-R score > 3 (intermediate risk, high risk, very high risk);
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
6. complete case information could be obtained.

Exclusion Criteria:

1. patients who did not meet the inclusion criteria;
2. inability to obtain complete case information or to follow protocol steps or follow up on time;
3. other conditions considered by the investigators to be unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older with newly diagnosed myelodysplastic agenda syndrome (MDS)and chronic myelomonocytic leukemia (CMML)according to the 2016WHO or 2022 WHO criteria
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | After the first cycles treatment（Day1, Month2)
  CR+mCR+PR+HI

SECONDARY OUTCOMES:
IWG2023 Composite response rate | After the first cycles treatment（Day1, Month2 )
  CR+CR-L+CRh+CRequ
overall survival | through study completion, an average of 1 year
  Refers to the time from the start of treatment to the patient's death or last follow-up.
Blood transfusion dependence | through study completion, an average of 1 year
  Change in proportion of transfusion dependence from the start of treatment
adaverse event rate | Up to 1 years after the last subject enrolled.
  Grade 3-4 adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No